CLINICAL TRIAL: NCT03940417
Title: Cumulative Summation Analysis of Learning Curve for Robot-Assisted Gastrectomy in Gastric Cancer
Brief Title: Learning Curve for Robot-Assisted Gastrectomy in Gastric Cancer
Acronym: LCFRAGIGC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2019LSK-005
Record Dates: First submitted 2018-11-18; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2018-11

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators prospectively collected the clinical data of Da Vinci robot-assisted radical gastrectomy patients conducted by the same group of physicians from October 2017 to October 2018. The learning curve of the surgery was analyzed with the moving average method and the cumulative sum analysis (CUSUM). The short-term efficacy was then validated by comparing the perioperative and pathologic outcomes of patients in the two stages of the learning curve.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients were 18-90 years old
* 2. Patients with a documented diagnosis of gastric adenocarcinoma
* 3. patients were scheduled to undergo minimally invasive gastric cancer surgery
* 4.patients with no preoperative evidence of serosal invasion or extraperigastric lymph node metastasis on preoperative computed tomography scans, upper endoscopy, and endoscopic ultrasound

Exclusion Criteria:

* 1. Patients with neoadjuvant treatment
* 2. Patients procedure concurrent with the gastrectomy
* 3.Patients with palliative surgery
* 4. Patients with the contraindications for general anesthesia
* 5. Patients were pregnant or mentally incompetent
* 6. Patients with serious systemic comorbidities, such as severe heart failure, respiratory failure, uncontrolled hypertension

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients were scheduled to undergo minimally invasive gastric cancer surgery and meet the above conditions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Operation time,min | 1 week
  The surgeon begins the operation until the incision is closed
Docking time,min | 1 week
  From the skin cutting through the observation hole to the robot moving to the designated position, the lens and the instrument arm enter the abdominal cavity and prepare for this period

SECONDARY OUTCOMES:
Evaluated blood loss ,ml | 1 week
  The amount of bleeding in the suction device plus the amount of bleeding dipped in the gauze
Number of retrieved lymph nodes | 1 week
  Refer to the postoperative pathology report
Day of ﬁrst ﬂatus,day | 2 week
Day of ﬁrst ﬂuid diet,day | 2 week
the rate of postoperative complications | 30 days after the operation
  Postoperative complications included infectious complications, intra-abdominal/intraluminal bleeding, gastric stasis and leakage
postoperative hospital stay, days | 30 days after the operation
  Length of postoperative hospital stay
cost | 30 days after the operation
  total cost in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi, China